CLINICAL TRIAL: NCT02168712
Title: Interval Versus Continuous Exercise Training on Functional Capacity and Quality of Life in Patients With Coronary Artery Disease: a Randomized Clinical Trial
Brief Title: Interval Versus Continuous Training on Functional Capacity and Quality of Life in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Responsible Party: Principal Investigator, KOLDO VILLELABEITIA JAUREGUIZAR, Chief of Rehabilitation Department, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EO31/2013-HIE
Record Dates: First submitted 2014-06-16; First posted 2014-06-20 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Heart Disease; Interval exercise training; Continuous exercise training; Quality of life; Safety
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate continuous exercise training (Active Comparator): Moderate intensity continuous exercise training
  Interventions: Other: Moderate continuous exercise training
- Interval exercise training (Experimental): High intensity interval exercise training
  Interventions: Other: Interval exercise training

INTERVENTIONS:
Other: Moderate continuous exercise training
  Arms: Moderate continuous exercise training
Other: Interval exercise training
  Arms: Interval exercise training

SUMMARY:
Exercise therapy increase functional capacity improving the morbidity and mortality of patients with cardiovascular disease. Moderate continuous training is the best established training modality for this patients. However, a body of evidence has begun to emerge demonstrating that high intensity interval training obtained better results in terms of morbidity and mortality.

The purpose of this randomized clinical trial was to determine the effect of two types of exercise training: moderate continuous training vs high interval training on functional capacity and quality of life as well as verify the safety in its application.

We included 72 patients with coronary artery disease by assigning one of the training modality for 8 weeks. We analyzed cyclo-ergo-spirometry data, aspect related to quality of life as well as a record of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Coronary heart Disease, with functional class II-III according to New York Heart Association classification system.
* At least 4 weeks from acute cardiac event, percutaneous or surgery revascularization.
* Optimized medical treatment in adequate doses ( betablockers, ACE inhibitors, ARA II, statins and antiplatelet drugs)
* Age > 18 years old.
* Willing to participate and sign an informed consent form

Exclusion Criteria:

* Residual ischemia waiting for revascularization.
* Any cardiac event for the last 4 weeks
* Abnormal Ergometry with hemodynamic or clinically significant arrhythmias during the procedure.
* History of severe ventricular arrhythmia
* Uncontrolled glycaemia or blood pressure
* Moderate to severe Chronic Pulmonary Obstructive Disease
* Osteomuscular and/or mental disorder that hampers an adequate adherence to the intervention program
* Other vascular diseases: rheumatologic/ autoimmune disorders, thrombopathies, hemophilia.
* Active oncologic disease.
* Treatment with corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Impact on functional capacity | 2 months
  Basal and peak oxygen consumption values will be measured.

SECONDARY OUTCOMES:
quality of life | 2 months
  Quality of life will be compared between the two arms with one generic questionnaire (SF-36) and one ischemic heart disease specific questionnaire (MacNew)

OTHER OUTCOMES:
Incidence of Adverse Events | 2 months
  The incidence of cardiovascular adverse events in each group will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infanta Elena, Valdemoro, Madrid, Spain